CLINICAL TRIAL: NCT07405983
Title: Effectiveness and Safety of the TOUCH® CMC 1 Prosthesis, Post-Approval Study
Brief Title: TOUCH® CMC 1 New Enrollment US Study
Acronym: PAS002
Status: Not yet recruiting | Type: Observational
Sponsor: Keri Medical SA (Industry)
Collaborators: MCRA (an IQVIA business) (Unknown)
Responsible Party: Sponsor
Other Study IDs: TOUCH® CMC 1 New Enrollment US
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis Thumb; Thumb Carpometacarpal Joint Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- TOUCH® CMC 1 Prosthesis
  Interventions: Device: TOUCH® CMC 1 Prosthesis

INTERVENTIONS:
Device: TOUCH® CMC 1 Prosthesis — The TOUCH® CMC 1 Prosthesis is a commercially available thumb joint implant which is made up of three modular components:
  1. TOUCH Cup: a stainless steel trapezial implant (cup) with a dual coating of plasma sprayed titanium and hydroxyapatite; TOUCH Cup is available in two options: Spherical and Conical
  2. TOUCH Liner and Neck: a junction implant (neck) topped with a liner pre-assembled to stainless steel neck
  3. TOUCH Stem: a titanium alloy metacarpal implant (stem) with a dual coating of plasma sprayed titanium and hydroxyapatite

SUMMARY:
The purpose of this study is to meet a PMA (P240020) condition of approval of the TOUCH® CMC 1 Prosthesis to evaluate the effectiveness and safety of the prosthesis in the United States (US) population. The device performance in newly enrolled US patients implanted by US surgeons will be compared to device performance observed within the outside the US (OUS) premarket cohort.

DETAILED DESCRIPTION:
TOUCH® CMC 1 (Carpometacarpal) Prosthesis is a cementless, ball-and-socket dual-mobility, total CMC1 joint replacement prosthesis, designed to treat osteoarthritis of the base of the thumb. The TOUCH® CMC 1 Prosthesis was approved by FDA (P240020) on July 10, 2025. Continued approval of the premarket approval application (PMA) is contingent upon the submission of periodic reports (Annual Report), required under 21 CFR 814.84. In order to provide continued reasonable assurance of the safety and effectiveness of the PMA device, data from this post-approval study must be submitted to FDA in a PMA Post Approval Study Report per the requirements set forth in the approval.

ELIGIBILITY:
Inclusion Criteria:

1. Patient requiring 1st carpometacarpal (CMC) primary total joint replacement (arthroplasty) to surgically treat symptomatic Eaton-Littler Stage II or III osteoarthritis (OA)
2. Adult (≥ 22 years of age) at the time of enrollment
3. Willing and able to sign the study Informed Consent

Exclusion Criteria:

1. Acute or chronic infections, local or systemic
2. Muscular, neurological, or vascular severe deficiency affecting the joint
3. Inadequate bone quality or quantity preventing the implant fixation
4. Bones dimensions incompatible with implant sizes
5. Patients who are allergic to the product's materials
6. Any concomitant disorder that may affect the function of the implant (e.g., osteoarthritis of the wrist)
7. Skeletally immature (i.e., pediatric population, <22 years of age)
8. Pregnant or nursing women
9. Patients with contraindications to surgery in general
10. Patients with an intellectual disability who cannot follow the instructions of their surgeon.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in this study will be recruited from the investigators' standard patient populations. All patients presenting with osteoarthritis of the 1st carpometacarpal joint will be evaluated for study participation based on the inclusion/exclusion criteria. Subjects must meet all of the following inclusion criteria and none of the exclusion criteria. The investigator maintains exclusive responsibility for the inclusion and exclusion of any potential study participant.
Sampling Method: Non-Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-11 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Composite Success | 24 Months/2 Years
  1. Improvement of pain: A clinically meaningful improvement in pain during activities defined as a decrease in the Numerical Rating Scale (NRS) pain score of ≥ 30% on a 10-point scale.
  2. Maintenance or improvement in function: defined by key pinch strength, which is ≥ 85% of the subject's pre-operative key pinch strength.
  3. Safety: success is defined as freedom from:
     * Subsequent surgical interventions (SSI) (i.e., reoperation, revision, removal of any study component, or supplemental fixations) on the study carpometacarpal joint, or
     * Serious, device- or procedure-related adverse events

IPD SHARING:
Plan to Share IPD: Undecided